CLINICAL TRIAL: NCT02674542
Title: Family Planning Intentions and Practices Among Women Who Have Experienced a Poor Obstetric Outcome: a Qualitative Study
Brief Title: Family Planning Intentions and Practices Among Women With Poor Obstetric Outcome
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: UNCPM 21416
Record Dates: First submitted 2016-01-22; First posted 2016-02-04 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Stillbirth
Keywords: Family planning; Birth spacing
MeSH Terms: conditions — Stillbirth | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: In-depth interviews — 1. Future family planning intentions and beliefs
  2. Family planning experiences and beliefs:
  3. Feasibility and acceptability of birth spacing promotion for women who experienced a still birth or early neonatal demise
Other: Focus Group — 1. Future family planning intentions and beliefs
  2. Family planning experiences and beliefs:
  3. Feasibility and acceptability of birth spacing promotion for women who have experienced a stillbirth or early neonatal demise

SUMMARY:
Women who have experienced a stillbirth or neonatal death are at higher risk of repeated poor neonatal outcomes if they have short interpregnancy intervals. Understanding the attitudes surrounding future fertility and contraception in this population is critical to propose socially and culturally acceptable interventions to address an unmet need for family planning.

Participants: Women who have experienced a stillbirth or early neonatal death will be recruited from the postnatal ward of Bwaila Maternity Hospital in Lilongwe, Malawi.

Procedures (methods): This will be a qualitative study using 20 in-depth interviews and four focus group discussions of up to 10 women each.

DETAILED DESCRIPTION:
The investigators propose a qualitative study of up to 60 women who have experienced a stillbirth or early neonatal death. This will be a qualitative study using 20 in-depth interviews and four focus group discussions of up to 10 women each. In-depth interviews will be conducted in Chichewa in a private room either within the participants' homes or in another private location determined by the participant.

Each interview will take approximately 60-90 minutes to complete. The focus group discussions will be conducted in a private room in a health facility with 6-10 participants. These will take approximately 90-120 minutes to complete. Interviews and the focus group discussion will be audio-recorded, transcribed, and translated to English. If a participant is found to be eligible, she will be invited to participate in the study. After the investigators complete the in-depth interviews, the investigators will analyze the data and modify our focus group discussion guide as needed to integrate new themes that may have emerged during the individual interviews. The investigators will recruit 6-10 women per focus group (24 to 40 total) from the same hospital that were used to recruit for the individual interviews.

The investigators will search for recurrent patterns and themes in data and for ideas that help to explain the presence of these patterns. The data collection and analysis process is designed to be iterative, such that the investigators will be reviewing data as it is collected and adjusting the data collection instrument to reflect new themes that emerge during the data collection process. All interviews will be audio-recorded, transcribed, translated, coded and computerized for analysis.

ELIGIBILITY:
Inclusion criteria:

1. Current admission to the postpartum ward at Bwaila Hospital,
2. Women who have delivered a stillborn fetus over 28 weeks gestation or with a birthweight >1000 g or experienced a neonatal demise of a liveborn infant, weighing >1000 g in the first 7 days of life,
3. Ability to speak Chichewa or English fluently, and
4. Age 18-45 years old.

Exclusion criteria:

* Not willing to be audio-recorded
* Have not experienced stillbirth or early neonatal death

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 60 women who have experienced a stillbirth or early neonatal death. Study participants will be recruited from the postnatal wards at Bwaila Maternity Hospital in Lilongwe, Malawi.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Attitudes surrounding future fertility, birth spacing, family size, and contraception | 1 year
  The investigators expect that the in-depth interviews and focus groups will allow them to better understand the family planning intentions and practices of women who have experienced a stillbirth or early neonatal demise.

SECONDARY OUTCOMES:
Discovering feasible and acceptable interventions to promote birth spacing and family planning among women who have experienced a poor obstetric outcome | 1 year
  The investigators will ask women who have experienced a stillbirth or neonatal demise questions about a variety of potential interventions to assist women with birth spacing and elicit their ideas on acceptable interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Kopp, MD, MPH, Principal Investigator — UNC-CH
Locations (1):
- UNC Project, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bula A, Kopp DM, Maman S, Chinula L, Tsidya M, Tang JH. Family planning knowledge, experiences and reproductive desires among women who had experienced a poor obstetric outcome in Lilongwe Malawi: a qualitative study. Contracept Reprod Med. 2018 Oct 17;3:22. doi: 10.1186/s40834-018-0075-8. eCollection 2018. PMID 30349736
- [Derived] Kopp DM, Bula A, Maman S, Chinula L, Tsidya M, Mwale M, Tang JH. Influences on birth spacing intentions and desired interventions among women who have experienced a poor obstetric outcome in Lilongwe Malawi: a qualitative study. BMC Pregnancy Childbirth. 2018 May 31;18(1):197. doi: 10.1186/s12884-018-1835-9. PMID 29855296